CLINICAL TRIAL: NCT00198432
Title: Randomized Phase II Study Evaluating an Induction Chemotherapy Followed by a Concomitant Chemoradiotherapy and a Concomitant Chemoradiotherapy Followed by a Consolidation Chemotherapy Among Patients With NSCLC Stage III Not Resectable
Brief Title: Chemoradiotherapy of NSCLC Stage IIIB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Collaborators: Bristol-Myers Squibb (Industry); Pierre Fabre Laboratories (Industry); Ligue contre le cancer, France (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-0201
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: NSCLC Stage IIIB; Concomitant Radiochemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Vinorelbine; Cisplatin

INTERVENTIONS:
Drug: Paclitaxel, vinorelbine, cisplatin

SUMMARY:
To evaluate the best timing of the concomitant chemoradiotherapy among patients with NSCLC stage III not resectable treated by concomitant chemo-radiotherapy, either preceded by a induction chemotherapy, or followed by a consolidation chemotherapy.

DETAILED DESCRIPTION:
Chemotherapy:

C = Cisplatine : 80 mg/m² P = Paclitaxel : 200 mg/m² N = Vinorelbine : 15 mg/m²

Radiotherapy:

66 Gy with 33 fractions (2 Gy/fraction, 1 fraction/day, 6,5 weeks) High energy Photons X (>= 9MV)

ELIGIBILITY:
Inclusion Criteria:

* NSCLC stage IIIA N2 or IIIB not resectable, except N3 sus-clavicular, nor reached pleural
* PS = 0 or 1
* Possibility of including all the targets in only one exposure field
* Slimming < 10% of the weight of the body
* Functions hepatic, renal and hematologic normal
* VEMS >40% and PaO2 >60 mmHg
* written and signed informed consent

Exclusion criteria :

- NSCLC stage IV or wet-IIIB

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2002-03; Study Completion 2006-12

PRIMARY OUTCOMES:
Objective response rate

SECONDARY OUTCOMES:
Overall survival
Time to progression
Relapse rate (local control)
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fournel, Dr, Principal Investigator — Intergroupe Francophone de Cancerologie Thoracique
Locations (1):
- CHU Saint-Etienne Pneumologie, Saint-Etienne, France

REFERENCES:
- [Result] Fournel P, Vergnenegre A, Robinet G, Lena H, Gervais R, Le Caer H, Souquet PJ, Chavaillon JM, Bozonnat MC, Daures JP, Chouaid C, Martel-Lafay I; GFPC and IFCT Team. Induction or consolidation chemotherapy for unresectable stage III non-small-cell lung cancer patients treated with concurrent chemoradiation: a randomised phase II trial GFPC - IFCT 02-01. Eur J Cancer. 2016 Jan;52:181-7. doi: 10.1016/j.ejca.2015.10.072. Epub 2015 Dec 12. PMID 26689864